CLINICAL TRIAL: NCT02905591
Title: A Phase 2 Trial of Pharmacological Ascorbate With Concurrent Chemotherapy and Radiation Therapy for Non-small Cell Lung Cancer
Brief Title: A Phase 2 Study Adding Ascorbate to Chemotherapy and Radiation Therapy for NSCLC
Acronym: XACT-LUNG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Joseph J. Cullen, MD, FACS (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Holden Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Bryan Allen, Assistant Professor, Department of Radiation Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201712770; 3P30CA086862 (NIH); 5U01CA140206 (NIH); 1P01CA217797-01A1 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Nonsmall Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; NSCLC
Keywords: pharmacological ascorbate; ascorbic acid; radiation; chemotherapy; carboplatin; paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated; Paclitaxel; Taxes; Carboplatin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ChemoRT + Ascorbate (Experimental): Radiation therapy, intravenous paclitaxel, intravenous carboplatin, intravenous ascorbic acid (pharmacological ascorbate)
  Interventions: Drug: Radiation Therapy; Drug: Paclitaxel; Drug: Carboplatin; Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Radiation Therapy — Conformal radiation administered daily, Monday through Friday Total dose is 60 Gray (Gy) and is delivered in 2 Gy fractions. One fraction is delivered daily for a total of 30 fractions in 30 days
  Other Names: external beam radiation therapy (EBRT); intensity modulated radiation therapy (IMRT); Volumetric Arc Therapy (VMAT); XRT
Drug: Paclitaxel — Administered intravenously (IV) Given the same day as carboplatin, but given before the carboplatin is administered
  * the dose is 45 mg/m2 (standard dose)
  * Administered weekly
  * 6 to 7 weeks of therapy, depending on when radiation starts
  * Standardized dose reductions are used
  Other Names: Nov-Onxol; Onxol; Paclitaxel Novaplus; Taxol
Drug: Carboplatin — Administered intravenously (IV) GIven the same day as paclitaxel, immediately after the paclitaxel infusion is done.
  * Prescribed at area-under-the-curve (AUC) = 2 using the Cockroft-Gault formula (standard)
  * Administered weekly
  * 6 to 7 weeks of therapy, depending on when radiation starts
  * Standard dose reductions are used
  Other Names: NovaPlus CARBOplatin; Amerinet Choice Carboplatin; Paraplatin; Paraplatin NovaPlus
Drug: Ascorbic Acid — Administered intravenously
  * 75 grams per infusion; each infusion is about 2 hours
  * 3 infusion per calendar week
  * The infusion is actively running for at least 20 minutes when radiation begins
  * May be given while chemotherapy is delayed due to low counts
  * Dose reductions are not used
  * Given for 6 to 7 weeks, depending on when radiation starts
  Other Names: Ascorbate; Vitamin C; Pharmacological ascorbate

SUMMARY:
This clinical trial evaluates adding high-dose ascorbate (vitamin C) to a standard therapy for non-small cell lung cancer. The standard therapy is radiation therapy combined with carboplatin and paclitaxel (types of chemotherapy). All subjects will receive high-dose ascorbate in addition to the standard therapy.

DETAILED DESCRIPTION:
For selected stages of non-small cell lung cancer (NSCLC), standard treatment involves radiation therapy and chemotherapy. The chemotherapy regimen typically used is paclitaxel and carboplatin. Both of these chemotherapeutic drugs are administered intravenously, using a vein in the arm. Radiation is administered using a machine external to the body (usually a linear accelerator). After combined therapy, NSCLC patients receive 2 extra cycles of chemotherapy, called "consolidation chemotherapy."

This study adds 75 grams of ascorbate (vitamin C, sometimes called pharmacological ascorbate because the dose is so high) at specific timepoints in the therapy. The ascorbate is administered intravenously - through a vein in your arm.

Participants will:

* receive 75 grams of intravenous ascorbate 3 times per calendar week while they are receiving radiation therapy. The IV will be running while the radiation therapy is administered.
* undergo imaging which is standard for their cancer and therapy. This can include CT scans, PET scans, and X-rays.
* provide blood samples to determine the biological effects, if any, the ascorbate has on the body during therapy

This active therapy portion lasts for about 10 to 12 weeks. After that is done, participants go back to standard follow-up for their cancer and any additional therapy their doctors believe they need.

However, it is very important the investigators remain in contact with participants; they will have life-long follow-up for this study.

ELIGIBILITY:
Inclusion Criteria:

Note: patients who have a small pleural effusion that is too small to safety tap and is not visible on a chest x-ray are still eligible

* Pathologic diagnosis (i.e., cell sample, biopsy, tissue swap, bronchoscopy) of non-small cell lung cancer.
* Recommended to receive carboplatin & paclitaxel with radiation therapy as a treatment
* Tumor or metastatic disease must measure at least 1 cm using a CT scan (CAT scan)
* Physician determined the patient is healthy enough for chemotherapy and radiation therapy
* At least part of the lung cancer must be viewable and measurable by CT or MRI
* A platelet count of at least 100,000 cells per mililiter
* A creatinine level of less than 1 1/2 times the upper limit of normal for the local lab test, or, a creatinine clearance of at least 60 mL/(min*1.73m2)
* Not pregnant, and commit to using birth control during the study

Exclusion Criteria:

* Exudative pleural effusion
* Recurrent non-small cell lung cancer
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients actively receiving insulin or patients whose doctors have recommended current insulin use
* Patients requiring daily finger-stick blood glucose measurements
* Patients who are on the following drugs and cannot have a substitution or who decline the substitution:

  * warfarin
  * flecainide
  * methadone
  * amphetamines
  * quinidine
  * chlorpropamide
* Prior radiation therapy that would result in a field overlap
* Enrolled in another therapeutic clinical trial
* Uncontrolled, intercurrent illness
* Lactating women
* HIV positive individuals undergoing therapy due to known drug:drug interaction between antiretroviral drugs and high-dose ascorbate therapy

If all the above are met, the potential participant will receive a 15 gram challenge dose of ascorbate via intravenous infusion. This is the final screening procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2025-07-17 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression rate at completion of radiation and chemotherapy | 3 to 4 weeks after last radiation treatment
  Tumor measurement from CT scan, using the RECIST criteria to define progression

SECONDARY OUTCOMES:
Tumor response | Every six months for up to 20 years post-treatment
  From radiation day 1 to documented disease progression as described by RECIST criteria. Results are provided in nominal categories (CR, PR, SD, PD) as per RECIST.
Progression free survival (PFS) | Every six months for up to 20 years post-treatment
  Time, measured in days, it takes for disease to progress, where disease progression is defined by the RECIST criteria (v1.1). Timeframe is from radiation day 1 to date of disease progression
Overall survival (OS) | Every three months for up to 20 years post-treatment
  Time, measured in months, from start of radiation to death from any cause.
Adverse event frequency and categorization | Weekly for the first 7 weeks, then monthly for 3 months, then every 6 months through 2 years post-treatment
  Categorize and quantify adverse events using the Common Terminology Criteria for Adverse Events (CTCAE, v 4) as follows:
  * Through radiation, weekly assessment of adverse events
  * Consolidation chemotherapy, assessment day 1 of each cycle
  * Post-treatment, every 6 months through 2 years post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Cullen, MD, FACS, Study Director — University of Iowa
Locations (1):
- Holden Comprehensive Cancer Cener, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared upon request in compliance with the IRB application and protocol.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon request.
Access Criteria: Contact the investigator or sub-investigator to initiate a request. A contract may be required between institutions. Data will be shared only from those participants who consented to sharing.

REFERENCES:
- [Background] Schoenfeld JD, Sibenaller ZA, Mapuskar KA, Wagner BA, Cramer-Morales KL, Furqan M, Sandhu S, Carlisle TL, Smith MC, Abu Hejleh T, Berg DJ, Zhang J, Keech J, Parekh KR, Bhatia S, Monga V, Bodeker KL, Ahmann L, Vollstedt S, Brown H, Shanahan Kauffman EP, Schall ME, Hohl RJ, Clamon GH, Greenlee JD, Howard MA, Schultz MK, Smith BJ, Riley DP, Domann FE, Cullen JJ, Buettner GR, Buatti JM, Spitz DR, Allen BG. O2⋅- and H2O2-Mediated Disruption of Fe Metabolism Causes the Differential Susceptibility of NSCLC and GBM Cancer Cells to Pharmacological Ascorbate. Cancer Cell. 2017 Apr 10;31(4):487-500.e8. doi: 10.1016/j.ccell.2017.02.018. Epub 2017 Mar 30. PMID 28366679

DOCUMENTS (1):
  • Informed Consent Form (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT02905591/ICF_001.pdf